CLINICAL TRIAL: NCT02779244
Title: Early Weight Bearing for Unstable Ankle Fractures Undergoing Operative Stabilization: Is It Safe and Does It Improve Outcomes?
Brief Title: Early Weight Bearing for Unstable Ankle Fractures Undergoing Operative Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-00720
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Ankle Fracture
Keywords: Orthopedic; Post-operative; Weight bearing; Range of motion
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Weight Bearing + Cam boot (Experimental)
  Interventions: Procedure: Early Weight bearing + Cam Boot
- Standard Treatment Cam boot (Active Comparator)
  Interventions: Procedure: Non-Weight Bearing + Cam Boot

INTERVENTIONS:
Procedure: Early Weight bearing + Cam Boot — Patients will be transitioned to weight bearing as tolerated in a cam boot.
  Arms: Early Weight Bearing + Cam boot
Procedure: Non-Weight Bearing + Cam Boot — Subject will be transitioned to non weight bearing cam boot, standard treatment.
  Arms: Standard Treatment Cam boot

SUMMARY:
The purpose of this randomized, controlled trial is to estimate the safety of early weight bearing on post ankle surgery.

Patients who are indicated to have surgery for unstable ankle fractures by an attending trauma physician will be consented for participation in the study. After surgery patients will be randomized to either weight bearing as tolerated at two weeks with a cam boot or non-weight bearing with a cam boot. Randomization will be performed by number allocation with odd numbers in the early weight bearing group and even numbers in the non-weight bearing group. The surgeon will be blinded to this until after the surgery. The patients will all be placed in a short leg cast post operative and made non-weight bearing for 2 weeks until sutures are removed which is current standard treatment. Both groups will be asked to initiate weight bearing at two weeks post operatively by wearing a cam boot that is non weight bearing in a cam boot, the latter being standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Operative unstable ankle fractures

Exclusion Criteria:

* Requirement of syndesmotic fixation
* Pilon fractures
* Open fractures
* Patients with diabetic neuropathy
* BMI>40
* Polytrauma patients
* Patients who are unable to comply with non-weight bearing
* Patients who are unable to follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Olerud Molander Ankle Score | 1 year
  The Olerud Molander score is scored between 0 - 100 as painless and functionally perfect ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmal Tejwan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States